CLINICAL TRIAL: NCT01392573
Title: A 26-week Randomised, Parallel Two-arm, Double-blind, Multi-centre, Multinational, Treat-to-target Trial Comparing Fixed Ratio Combination of Insulin Degludec and Liraglutide With Insulin Degludec in Subjects With Type 2 Diabetes
Brief Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec/Liraglutide and Insulin Degludec in Subjects With Type 2 Diabetes
Acronym: DUAL™ II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9068-3912; 2011-002336-72 (EudraCT Number); U1111-1121-4897 (Other: WHO)
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegLira + metformin (Experimental): IDegLira was injected subcutaneously once daily for 26 weeks.
  Interventions: Drug: insulin degludec/liraglutide
- IDeg + metformin (Experimental): IDeg was injected subcutaneously once daily for 26 weeks.
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec/liraglutide — IDeg/Lira treatment will be initiated and titrated (individually adjusted) twice weekly according to the mean self measured plasma glucose (SMPG) (fasting). IDegLira is injected subcutaneously (under the skin) once daily.
  Arms: IDegLira + metformin
Drug: insulin degludec — IDeg treatment will be initiated and titrated (individually adjusted) twice weekly according to the mean self measured plasma glucose (SMPG) (fasting). IDeg is injected subcutaneously (under the skin) once daily.
  Arms: IDeg + metformin

SUMMARY:
This trial is conducted in Asia, Europe and the United States of America (USA). The aim of this trial is to compare the efficacy and safety of insulin degludec/liraglutide (IDegLira) and insulin degludec (IDeg) in subjects with type 2 diabetes. Subjects continue their pre-trial treatment with metformin throughout the entire trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* HbA1c (glycosylated haemoglobin) 7.5-10.0% (both inclusive)
* Subjects on stable daily doses for at least 90 days prior to trial start of: Basal insulin (total daily basal insulin dose within the range of 20-40U in combination with: metformin (1500 mg or more or max. tolerated dose) or metformin (1500 mg or more or max. tolerated dose) and SU (sulfonylurea) (equal to or more than half of the max. approved dose according to local label) or metformin and glinides (equal to or more than half of the max. approved dose according to local label)
* BMI (Body Mass Index) more than or equal to 27 kg/m^2

Exclusion Criteria:

* Treatment with glucagon like peptide-1 (GLP-1) receptor agonists (e.g. exenatide, liraglutide), dipeptidyl peptidase 4 (DPP-4) inhibitors and/or thiazolidinediones within 90 days prior to trial start
* Impaired liver function
* Impaired renal function
* Screening calcitonin equal to or above 50 ng/l
* Subjects with personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN 2)
* Cardiac disorder defined as: congestive heart failure (NYHA class III-IV), diagnosis of unstable angina pectoris, cerebral stroke and/or myocardial infarction within the last 52 weeks prior to trial start and/or planned coronary, carotid or peripheral artery revascularisation procedures
* Severe uncontrolled treated or untreated hypertension (systolic blood pressure equal to or above 180 mm Hg or diastolic blood pressure equal to or above 100 mm Hg)
* Acute treatment required proliferative retinopathy or maculopathy (macular oedema) according to physician's opinion
* History of chronic pancreatitis or idiopathic acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2011-11-28 (Actual); Primary Completion 2012-10-01 (Actual); Study Completion 2012-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (79):
- United States (52):
  - Novo Nordisk Investigational Site, Huntsville, Alabama
  - Novo Nordisk Investigational Site, Vestavia Hills, Alabama
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Arlington Heights, Illinois
  - Novo Nordisk Investigational Site, Avon, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, New Albany, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Methuen, Massachusetts
  - Novo Nordisk Investigational Site, North Dartmouth, Massachusetts
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Saint Charles, Missouri
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Smithtown, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Hickory, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
- Bulgaria (6):
  - Novo Nordisk Investigational Site, Burgas
  - Novo Nordisk Investigational Site, Haskovo
  - Novo Nordisk Investigational Site, Lukovit
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sofia
- Denmark (3):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Gentofte Municipality
  - Novo Nordisk Investigational Site, Hellerup
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Szombathely
- India (5):
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Dhantoli, Nagpur
- Slovenia (3):
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Ljubljana
  - Novo Nordisk Investigational Site, Novo Mesto
- Switzerland (6):
  - Novo Nordisk Investigational Site, Basel
  - Novo Nordisk Investigational Site, Bern
  - Novo Nordisk Investigational Site, Interlaken-Unterseen
  - Novo Nordisk Investigational Site, Lausanne
  - Novo Nordisk Investigational Site, Lucerne
  - Novo Nordisk Investigational Site, Sankt Gallen

REFERENCES:
- [Background] Khunti K, Mohan V, Jain SM, Boesgaard TW, Begtrup K, Sethi B. Efficacy and Safety of IDegLira in Participants with Type 2 Diabetes in India Uncontrolled on Oral Antidiabetic Drugs and Basal Insulin: Data from the DUAL Clinical Trial Program. Diabetes Ther. 2017 Jun;8(3):673-682. doi: 10.1007/s13300-017-0252-9. Epub 2017 Mar 22. PMID 28332144
- [Background] Ericsson A, Lundqvist A. Cost Effectiveness of Insulin Degludec Plus Liraglutide (IDegLira) in a Fixed Combination for Uncontrolled Type 2 Diabetes Mellitus in Sweden. Appl Health Econ Health Policy. 2017 Apr;15(2):237-248. doi: 10.1007/s40258-016-0301-y. PMID 28063135
- [Result] Buse JB, Vilsboll T, Thurman J, Blevins TC, Langbakke IH, Bottcher SG, Rodbard HW; NN9068-3912 (DUAL-II) Trial Investigators. Contribution of liraglutide in the fixed-ratio combination of insulin degludec and liraglutide (IDegLira). Diabetes Care. 2014 Nov;37(11):2926-33. doi: 10.2337/dc14-0785. Epub 2014 Aug 11. PMID 25114296
- [Result] Vilsboll T, Vora J, Jarlov H, Kvist K, Blonde L. Type 2 Diabetes Patients Reach Target Glycemic Control Faster Using IDegLira than Either Insulin Degludec or Liraglutide Given Alone. Clin Drug Investig. 2016 Apr;36(4):293-303. doi: 10.1007/s40261-016-0376-0. PMID 26894800
- [Result] King AB, Philis-Tsimikas A, Kilpatrick ES, Langbakke IH, Begtrup K, Vilsboll T. A Fixed Ratio Combination of Insulin Degludec and Liraglutide (IDegLira) Reduces Glycemic Fluctuation and Brings More Patients with Type 2 Diabetes Within Blood Glucose Target Ranges. Diabetes Technol Ther. 2017 Apr;19(4):255-264. doi: 10.1089/dia.2016.0405. Epub 2017 Mar 10. PMID 28282219
- [Result] Lingvay I, Handelsman Y, Linjawi S, Vilsboll T, Halladin N, Ranc K, Liebl A. EFFICACY AND SAFETY OF IDEGLIRA IN OLDER PATIENTS WITH TYPE 2 DIABETES. Endocr Pract. 2019 Feb;25(2):144-155. doi: 10.4158/EP-2018-0284. Epub 2018 Nov 1. PMID 30383495
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 75 sites in 7 countries: Bulgaria (6), Switzerland (2), Denmark (3), Hungary (3), India (6), Slovenia (3), and the United States (52).
Groups:
- IDegLira: Insulin degludec/liraglutide (IDegLira) was injected subcutaneously (under the skin) once daily for 26 weeks in combination with metformin treatment. Metformin dose was maintained at the stable, pre-randomisation dose and frequency level. Treatment with IDegLira was initiated at 16 dose steps containing 16 units insulin degludec and 0.6 mg liraglutide. Dose adjustment of IDegLira was to be performed twice weekly based on the mean of three pre-breakfast self-monitored plasma glucose (SMPG) values measured on the day of titration and the two days prior to titration aiming at a fasting glycaemic target of 4.0-5.0 mmol/L.
- IDeg: Insulin degludec (IDeg) was injected subcutaneously (under the skin) once daily for 26 weeks. Metformin dose was maintained at the stable, pre-randomisation dose and frequency level. Treatment with IDeg was initiated with 16 units. Dose adjustment of IDeg was to be performed twice weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days (fasting glycaemic target of 4.0-5.0 mmol/L).
Period: Overall Study
Arm/Group | IDegLira | IDeg
Started | 207 | 206
Exposed | 207 | 206
Completed | 175 | 171
Not Completed | 32 | 35
Not completed — Adverse Event | 1 | 3
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal Criteria | 13 | 15
Not completed — Site closure | 8 | 7
Not completed — Unclassified | 9 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised subjects except 15 subjects (8 in IDegLira arm and 7 in IDeg arm) that were excluded due to site closure.
Groups:
- IDegLira: IDegLira was injected subcutaneously (under the skin) once daily for 26 weeks in combination with metformin treatment. Metformin dose was maintained at the stable, pre-randomisation dose and frequency level. Treatment with IDegLira was initiated at 16 dose steps containing 16 units insulin degludec and 0.6 mg liraglutide. Dose adjustment of IDegLira was to be performed twice weekly based on the mean of three pre-breakfast SMPG values measured on the day of titration and the two days prior to titration aiming at a fasting glycaemic target of 4.0-5.0 mmol/L.
- Total: Total of all reporting groups
Arm/Group | IDegLira | IDeg | Total
Number analyzed (Participants) | 199 | 199 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (8.9) | 57.5 (10.5) | 57.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 93 | 180
  Male | 112 | 106 | 218
HbA1c (glycosylated haemoglobin) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.7 (0.7) | 8.8 (0.7) | 8.8 (0.7)
Body Weight [Mean (Standard Deviation); unit: kg] | 95.4 (19.4) | 93.5 (20.0) | 94.5 (19.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Observed mean change from baseline in HbA1c after 26 Weeks of treatment.
Time Frame: Week 0, week 26
Population: Full analysis set. Missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegLira | IDeg
Number analyzed (Participants) | 199 | 199
percentage of glycosylated haemoglobin | -1.90 (1.09) | -0.89 (1.18)
Statistical Analysis 1: Comparison: IDegLira vs IDeg; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with treatment, country and previous antidiabetic treatment as fixed effects and baseline HbA1c value as covariate; Treatment contrast = -1.05, 95% CI 2-sided [-1.25 to -0.84]

2. Secondary Outcome: Change in Body Weight
Description: Observed mean change from baseline in body weight after 26 Weeks of treatment.
Time Frame: Week 0, week 26
Population: Full analysis set. Missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDegLira | IDeg
Number analyzed (Participants) | 199 | 199
kg | -2.7 (3.7) | 0.0 (3.4)

ADVERSE EVENTS:
Time Frame: Adverse events were captured from the time of consent untill 26 weeks of treatment, and were followed-up for 7 days after the final visit (upto overall 27 weeks).
Description: Safety analysis set included all subjects receiving at least one dose of the investigational product or comparator except 15 subjects (8 in IDegLira arm and 7 in IDeg arm) that were excluded due to site closure. Subjects in the safety analysis set contributed to the evaluation "as treated".
Arm/Group | IDegLira | IDeg
Serious Adverse Events (participants affected / at risk) | 7/199 | 11/199
Other Adverse Events (participants affected / at risk) | 45/199 | 29/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=199) | IDeg (N=199)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegLira (N=199) | IDeg (N=199)
Diarrhoea (Gastrointestinal disorders) | 13 (21) | 7 (8)
Nausea (Gastrointestinal disorders) | 13 (20) | 7 (7)
Nasopharyngitis (Infections and infestations) | 5 (5) | 12 (14)
Lipase increased (Investigations) | 12 (12) | 7 (7)
Headache (Nervous system disorders) | 12 (23) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.